CLINICAL TRIAL: NCT04705857
Title: Comparative Study of Gene-activated Bone Substitute Based on Octacalcium Phosphate and Plasmid DNA Encoding VEGFA Gene Mixed With Autobone and Bone Autograft From Iliac Crest in Treatment of Long Bone Nonunions With Bone Loss: an Open-label Randomized Controlled Trial
Brief Title: Comparative Study of Gene-activated Bone Substitute and Autobone in Treatment of Long Bone Nonunions
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Histograft Co., Ltd. (Industry)
Collaborators: S. M. Kirov Military Medical Academy of the Ministry of Defense of the Russian Federation (Other)
Responsible Party: Sponsor
Other Study IDs: Histograft-NONUNION-1.0
Record Dates: First submitted 2021-01-11; First posted 2021-01-12 (Actual); Last update posted 2021-01-13 (Actual); Status verified 2020-08

CONDITIONS: Non Union Fracture; Non-Union of Ankle Joint Without Infection
Keywords: nonunion; gene-activated matrix; bone grafting; bone substitute; VEGF; octacalcium phosphate
MeSH Terms: conditions — Fractures, Ununited

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- test group: bone reconstructive surgery with the use of "Histograft" bone substitute (gene-activated matrix based on octacalcium phosphate and plasmid DNA encoding VEGFA gene) mixed with shredded autobone (in a ratio of 50/50) harvested during the surgery
  Interventions: Combination Product: "Histograft", a bone substitute based on octacalcium phosphate (OCP) and plasmid DNA encoding VEGFA gene
- control group: bone reconstructive surgery with the use of shredded bone autograft harvested from iliac crest

INTERVENTIONS:
Combination Product: "Histograft", a bone substitute based on octacalcium phosphate (OCP) and plasmid DNA encoding VEGFA gene — gene-activated bone substitute in granular form, concentration of the plasmid DNA is 100 μg per 1.0 g of the OCP scaffold
  Groups: test group

SUMMARY:
The study is aimed to compare the effectiveness of "Histograft" bone substitute (gene-activated bone substitute based on octacalcium phosphate and plasmid DNA encoding VEGFA gene) mixed with shredded autobone and pure shredded auto bone harvested from iliac crest in treatment of patients with long bone nonunions

DETAILED DESCRIPTION:
An open-label randomized controlled clinical trial, two cohorts. Patients who met the inclusion criteria are planned to be enrolled into the trial. Upon enrollment, all patients will undergo screening, a set of clinical examination, instrumental investigations and laboratory tests, including CT of the affected bone with the assessment of nonunion.

All patients enrolled in the study will be subjected to bone reconstructive surgery with nonunion excision and bone grafting with either investigational bone substitute mixed with shredded autobone (in a ratio of 50/50) harvested during the surgery or pure shredded autobone from iliac crest.

The clinical study results will be evaluated at the time points of 1, 15, 45, 90, 180 days with clinical examination, instrumental investigations and laboratory tests. Control CT will be carried out for the primary outcome measure at 90, 180, 360 days after surgery.

ELIGIBILITY:
Inclusion Criteria:

* traumatic isolated closed or open Gustilo I and II, IIIA and IIIB humerus, tibial or femur diaphyseal or metaphysodiaphyseal fracture with a status of atrophic, oligotrophic or normotrophic non-union;
* signed voluntary informed consent

Exclusion Criteria:

* hypertrophic non-union;
* disability or unwillingness to give a voluntary informed consent or follow requirements of the clinical trial;
* segmental bone loss requiring specific therapy (bone transport, vascularized graft, large structural allograft, megaprosthesis, etc);
* other fractures causing interference with weight bearing;
* visceral injuries or diseases interfering with callus formation (severe cranioencephalic trauma, etc.);
* unrecovered vascular or neural injury;
* infection of any location and aetiology;
* pregnancy, breast feeding women and women who are of childbearing age and not practicing adequate birth control;
* malignant tumour (past history or concurrent disease);
* history of bone harvesting on iliac crest contraindicating new iliac crest bone graft harvesting or bone marrow collection;
* conditions limiting study compliance (e.g., dementia, psycho-neurological diseases, drug addiction, and alcoholism);
* medication affecting bone turnover (oral bisphosphonates, PTH, sodium fluoride, strontium ranelate, calcitonin, testosterone, systemic cortico- or anabolic steroids)

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients aged 18-70 with non-unions of long bones
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2022-08-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
Bone consolidation | 12 months
  Radiographic assessment of bone healing using REBORNE scale

SECONDARY OUTCOMES:
Adverse Events and Serious Adverse Events | 12 months
  Evaluation of the Adverse Events and Serious Adverse Events frequency
Ability to use the operated limb | 12 months
  Clinical assessment using DASH scale (for upper limb) or LEFS scale (for lower limb)
Pain level | 12 months
  Level of pain measured using Numeric Rating Scale

CONTACTS AND LOCATIONS:
Locations (1):
- S.M. Kirov Military Medical Academy, Department of Traumatology and Orthopaedics, Saint Petersburg, Russia

IPD SHARING:
Plan to Share IPD: Undecided
IPD could be shared through official depositories located on the clinical base official web site